CLINICAL TRIAL: NCT03945604
Title: A Phase Ib，Open-labeled, Multi-center, Dose-exploring Trial of SHR-1210 (Anti-PD-1 Antibody) in Combination With Apatinib and Fluzoparib in Subjects With Recurrent and Metastatic Triple Negative Breast Cancer
Brief Title: A Trial of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Apatinib and Fluzoparib in Patients With TNBC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-Ib-105
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; apatinib; fluzoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + Apatinib +Fluzoparib (Experimental): SHR-1210 will be administered as an intravenous infusion Apatinib tablets will be given orally Fluzoparib capsule will be given orally 28 days per cycle, until disease progression or unacceptable toxicity
  Interventions: Drug: SHR-1210 + Apatinib +Fluzoparib

INTERVENTIONS:
Drug: SHR-1210 + Apatinib +Fluzoparib — SHR-1210 will be administered as an intravenous infusion Apatinib tablets will be given orally Fluzoparib capsule will be given orally 28 days per cycle, until disease progression or unacceptable toxicity.
  Other Names: Treatment group ： PD-1 antibody SHR-1210 combination with apatinib and fluzoparib

SUMMARY:
The study is being conducted to evaluate the tolerability, safety and efficacy of SHR-1210 in combination with Apatinib and Fluzoparib in subjects with recurrent and metastatic triple negative breast cancer

DETAILED DESCRIPTION:
Drug: SHR-1210 + Apatinib +Fluzoparib SHR-1210 will be administered as an intravenous infusion, Apatinib tablets will be given orally, Fluzoparib capsule will be given orally 28 days per cycle, until disease progression or unacceptable toxicity.

Treatment group ： PD-1 antibody SHR-1210 combination with apatinib and fluzoparib

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent.
* Female aged ≥18 years old.
* Histologically diagnosed patients with recurrent and metastatic triple negative breast cancer.
* No more than 2-line chemotherapy failed at the stage of recurrence and metastasis .
* Patients who have been treated with platinum-based regimen at the stage of recurrence/metastasis need non-disease progression (non-pd)during treatment
* At least one measuring lesion that confirmed by RECIST v1.1 standard.
* The patients can swallow pills.
* Have a life expectancy of at least 12 weeks.
* The functions of vital organs meet protocal requirements.

Exclusion Criteria:

* Subjects had any history of active autoimmune disease .
* Subjects had previously been treated with anti-PD-1 and PD-L1 antibodies, or was known to be allergic to antibody drugs, or had previously been treated with apatinib, or had previously been treated with PARP inhibitors.
* Subjects have untreated central nervous system metastasis.
* History of hypertension and antihypertensive medications are not well controlled.
* Some clinical symptoms or diseases of the heart that are not well controlled.
* History of immunodeficiency including HIV-positive.
* Subjects had active infections.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female
Enrollment: 32 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | First cycle (28 days)
  Dose Limiting Toxicity

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | from the first drug administration to within 90 days for the last SHR-1210 dose
  AEs and SAEs
Overall Response Rate (ORR) | up to 12 months (approx) from the start of treatment
Duration of response (DoR) | up to 12 months (approx) from the start of treatment
Disease Control Rate | up to 12 months (approx) from the start of treatment
  DCR
Progression-Free-Survival | up to 12 months (approx) from the start of treatment
  PFS
12-months overall survival rate | From the start of treatment to 1 year
  12-months overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, PhD, Principal Investigator — Beijing Cancer Hosptial
Locations (1):
- Beijing Cancer Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang Q, Shao B, Tong Z, Ouyang Q, Wang Y, Xu G, Li S, Li H. A phase Ib study of camrelizumab in combination with apatinib and fuzuloparib in patients with recurrent or metastatic triple-negative breast cancer. BMC Med. 2022 Oct 3;20(1):321. doi: 10.1186/s12916-022-02527-6. PMID 36184642